CLINICAL TRIAL: NCT03361306
Title: LCI-HEM-MYE-CRD-002: A Phase II Study of Carfilzomib- Revlimid-Dexamethasone-Elotuzumab in Relapsed/Refractory Multiple Myeloma
Brief Title: LCI-HEM-MYE-CRD-002: Carfilzomib-Revlimid-Dexamethasone-Elotuzumab in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Bristol-Myers Squibb (Industry); Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-HEM-MYE-CRD-002; 00023493 (Other: Advarra IRB)
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Relapsed
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KRd-Elotuzumab (Experimental): Induction (4 28-day cycles):
  Carfilzomib (IV) @ 20 mg/m^2, Day 1 of Cycle 1; @ 56 mg/m^2, Day 8,15 of Cycle 1; @ 56 mg/m^2, Day 1,8,15 of Cycles 2-4
  Lenalidomide (Oral) @ 25 mg, once daily at bedtime on Days 1-21 of each cycle (Cycles 1-4)
  Dexamethasone @ 28 mg orally OR 8 mg IV, once weekly on Day 1,8,15,22 of Cycles 1-2; @28 mg orally OR 8 mg IV on Day 1 of Cycles 3-4
  Elotuzumab (IV) @ 10 mg/kg, once weekly on Day 1,8,15,22 of Cycles 1-2; @ 20 mg/kg on Day 1 of Cycles 3-4
  Maintenance (28-day cycles):
  Elotuzumab (IV) @ 20 mg/kg, Day 1 of each cycle (Cycles 1-n)
  Lenalidomide (Oral) @ 15 mg (or last tolerated dose if <15 mg), once daily at bedtime on Days 1-21 of each cycle (Cycles 1-n)
  Interventions: Drug: Elotuzumab

INTERVENTIONS:
Drug: Elotuzumab — Experimental
  Other Names: Empliciti

SUMMARY:
The study drug elotuzumab, has been clinically shown to be effective in treating relapsed/refractory MM in combination with either bortezomib, or lenalidomide and dexamethasone. Elotuzumab in combination with lenalidomide and dexamethasone is currently approved by the Food and Drug Administration (FDA) for the treatment of patients with multiple myeloma. Carfilzomib is also FDA approved for treating multiple myeloma and frequently given in combination with lenalidomide and dexamethasone for treatment of relapsed/refractory MM. Based on these findings, this study will look at how subjects with relapsed/refractory MM respond to a combination treatment with the following drugs: elotuzumab, carfilzomib, lenalidomide and dexamethasone. The combination of these four drugs is not FDA approved and is experimental.

DETAILED DESCRIPTION:
This single arm, open-label phase II study is designed with the primary objective of evaluating the efficacy of induction therapy comprised of 4 cycles of carfilzomib, lenalidomide, dexamethasone and elotuzumab (KRd+elotuzumab) in terms of very good partial response or better (VGPR+) in subjects with relapsed and/or refractory MM, and comparing to relevant historical controls. Post induction, all subjects will undergo disease evaluation for assessment of the primary endpoint. Maintenance therapy comprised of elotuzumab and lenalidomide (R+elotuzumab) will start directly after induction and continue until relapse or progression.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information signed by the subject or his/her legally authorized representative.
2. Age >= 18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 (see Appendix A, Section 18.1).
4. Documented history of relapsed and/or refractory multiple myeloma per IMWG 2016 criteria [22] as defined below (biochemical and/or clinical relapse per IMWG criteria); (NOTE: subjects refractory to bortezomib and/or lenalidomide are eligible; subjects who previously received carfilzomib are eligible provided they experienced a minimal response or better and relapsed >60 days after completion of treatment [see exclusion criteria #2]):

   1. Relapse is defined as progression of disease after an initial response to previous treatment, more than 6 months after discontinuation of treatment.
   2. Refractory is defined as lack of response to previous treatment, progression of disease during treatment, or progression of disease within 6 months of discontinuation of treatment.
5. Prior treatment with one line (and no more than one line) of systemic therapy for MM; NOTE: A new line of therapy is considered to start when a planned course of therapy is modified to include other treatment agents (alone or in combination) as a result of progressive disease (PD), relapse, or toxicity or when a planned period of observation off therapy is interrupted by a need for additional treatment for the disease. Induction therapy and stem cell transplant followed by planned maintenance therapy (provided there is no intervening PD) are considered to be a single line.
6. Subject must have recovered from any treatment-induced toxicities to ≤ grade 1 or baseline
7. Adequate washout from previous therapy:

   1. Prior chemotherapy is completed >3 weeks prior to day 1 of treatment (6 weeks for melphalan, nitrosoureas or monoclonal antibodies).
   2. Autologous transplant completed (referring to day of stem cell infusion) >12 weeks prior to day 1 of treatment; allogeneic transplant >16 weeks prior to day 1 of treatment.
   3. Prior radiotherapy completed at least 2 weeks prior to day 1 of treatment.
   4. Corticosteroid therapy at a dose equivalent to dexamethasone >4mg/day has been completed at least 2 weeks prior to day 1 of treatment.
8. Measurable disease defined as:

   1. Serum M-protein > 0.5 g/dL OR
   2. Urine M-protein ≥200 mg/24 h OR
   3. Involved free light chain (FLC) level ≥10 mg/dL provided serum FLC ratio is abnormal.
9. Demonstrate adequate organ function within 1 week of day 1 of treatment as defined in the table in Sec.tion 3.2 of protocol (#8)
10. Adequate cardiac function as defined by ≥45% Left Ventricular Ejection Fraction (LVEF) by ECHO or MUGA within 28 days prior to day 1 of treatment.
11. Females of childbearing potential (FCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to day 1 of treatment, and be willing to undergo serial serum or urine pregnancy testing. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause).
12. FCBP must be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) plus a second contraceptive method (considered acceptable [failure rate of >1% per year] or highly effective) from the time of informed consent until 6 months after the last protocol prescribed therapy has been discontinued. NOTE: estrogens may further increase the risk of thrombosis (beyond that associated with lenalidomide) and their use should be based on a benefit-risk decision. For the highly effective contraceptive method, a method with low user dependency is preferable but not required (see tables, adapted from:

    http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf).
13. Male subjects (even those who have had a vasectomy) who are sexually active with a FCBP must be willing to use latex or synthetic condoms from the time of informed consent until 180 days after the last protocol prescribed therapy has been discontinued. The FCBP partner should also consider contraception recommendations (see inclusion #11).
14. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

1. Discontinuation of previous lenalidomide, carfilzomib or dexamethasone due to intolerance.
2. If previously treated with carfilzomib, lack of response, progression during or relapsed within 60 days after completion of treatment.
3. Any infection, at the time of screening, requiring systemic therapy (i.e. involving IV antibiotics) (NOTE: at discretion of investigator, subjects with uncomplicated urinary tract infections may be eligible).
4. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study, and any female subject must agree not to donate eggs during the study and for 4 months after the last protocol prescribed therapy has been discontinued).
5. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, carcinoma of the prostate with a current PSA value of <0.5 ng/mL or other cancer for which the subject has completed treatment, been disease-free for at least five years, and is considered by Sponsor-Investigator to be at <30% risk of relapse, or on hormonal therapy for a history of either prostate cancer or breast cancer, provided that there has been no evidence of disease progression during the previous three years.
6. Non-secretory MM.
7. Active involvement of the central nervous system by MM.
8. Prior cardiovascular cerebrovascular accident with persistent neurological deficit.
9. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
10. Had major surgery within 4 weeks prior to day 1 of treatment.
11. Plasmapheresis within 4 weeks from day 1 of treatment.
12. Treatment with any investigational drug within 4 weeks prior to day 1 of treatment.
13. Uncontrolled clinically significant illness including, but not limited to, uncontrolled hypertension (as per the most updated Joint National Committee for the Management of Hypertension definitions), symptomatic congestive heart failure (as per New York Heart Association [NYHA] class III or IV [see Appendix C, Section 18.3], uncontrolled angina pectoris, myocardial infarction within the past 6 months, known or suspected amyloidosis, uncontrolled cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator, or any other condition (including laboratory abnormalities) that would, in the opinion of the Sponsor-Investigator, place the subject at unacceptable risk if he/she were to participate in the study.
14. Known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, elotuzumab or its excipients or known sensitivity to mammalian-derived products, carfilzomib or its excipients, lenalidomide or its excipients, or dexamethasone or its excipients.
15. Known human immunodeficiency virus (HIV) infection or active hepatitis A, B and/or C infection.

    1. Subjects with resolved HBV infection (i.e. subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Subjects who are PCR positive will be excluded. Exception: subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) and a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2025-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Bhutani, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhutani M, Foureau DM, Robinson M, Guo F, Fesenkova K, Atrash S, Paul B, Varga C, Friend R, Pineda-Roman M, Rigby K, Symanowski JT, Norek S, Tucker MR, Druhan LJ, Voorhees PM, Usmani SZ. A Clinical and Correlative Study of Elotuzumab, Carfilzomib, Lenalidomide, and Dexamethasone (Elo-KRd) for Lenalidomide Refractory Multiple Myeloma in First Relapse. Clin Lymphoma Myeloma Leuk. 2023 Jul;23(7):535-544.e1. doi: 10.1016/j.clml.2023.03.016. Epub 2023 Apr 7. PMID 37127471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KRd-Elotuzumab
Started | 15
Completed | 9
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | KRd-Elotuzumab
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 64 [46 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With VGPR or Better Response to Induction
Description: The primary endpoint is a binary variable determined for each subject indicating whether the subject achieved a very good partial response (VGPR), complete response (CR), or stringent complete response (sCR) to induction treatment with KRd-Elo, as defined by the IMWG 2016 response criteria. Per IMWG 2016 criteria, VGPR is defined as serum/urine M-protein detectable by immunofixation but not electrophoresis OR >= 90% reduction in serum M protein plus urine M-protein <100 mg/24 h. CR is defined as negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow aspirates. sCR is defined as CR plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry.
Time Frame: From enrollment to the disease response determined at the end of the induction part of regimen (4 cycles of KRd-Elo was planned, but some subjects progressed before the end of induction). The median length of induction was 16 weeks.
Population: The response evaluable population is defined as all subjects who initiate treatment with elotuzumab and who have measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | KRd-Elotuzumab
Number analyzed (Participants) | 15
Participants | 7
Statistical Analysis 1: Comparison: KRd-Elotuzumab; Test type: Superiority — Assuming the true VGPR+ rate is 40% under the null hypothesis, then this design will provide 90% power to detect a difference of 20% under the alternative hypothesis, assuming a one-sided alpha=0.10 significance level. For the originally planned enrollment of 40 subjects, if at least 21 subjects achieved VGPR or better to induction, the null hypothesis would be rejected; p = 0.390, Fisher Exact — This p-value is only based on partial enrollment on the study. As enrollment was halted early, this p-value is descriptive in nature and cannot determine the success/failure of the trial; Response Rate = 0.467, 95% CI 2-sided [0.213 to 0.734] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Number of Subjects With an Objective Response
Description: Objective response was determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of complete response (CR) or partial response (PR) as determined by IMWG 2016 response criteria.
Time Frame: From enrollment to best response while on study treatment; subjects remained on treatment until disease progression or death or unacceptable toxicity.
Reporting Status: Not Posted, anticipated posting 2026-02

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from treatment start date to the date of death from any cause. Subjects who are alive or lost to follow up at the time of the analysis will be censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described; assessed for approximately 5 years.
Reporting Status: Not Posted, anticipated posting 2026-02

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from treatment start date to first occurrence of either progressive disease (PD) or death. PD must be objectively determined per IMWG 2016 criteria, where progression date is date of last assessment that identified PD. If subject died without documented PD, progression date will be death date. For surviving subjects who do not have PD, PFS will be censored at the date of last disease assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, PFS will be censored at the date of last disease assessment prior to commencement of subsequent therapy. Subjects who have an initial PFS event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Time Frame: From treatment start date to date of progression/death, or censored as described; assessed for approximately 3 years.
Reporting Status: Not Posted, anticipated posting 2026-02

5. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP is defined as the duration of time from treatment start date to first occurrence of either progressive disease (PD) or death related to disease progression. PD must be objectively determined per IMWG 2016 criteria, where progression date is date of last assessment that identified PD. If a subject died for causes related to disease progression then progression date will be date of death. If a subject died for causes other than disease progression, TTP will be censored at the date of other cause mortality. For surviving subjects who do not have PD, TTP will be censored at the date of last disease assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, TTP will be censored at the date of last disease assessment prior to commencement of subsequent therapy. Subjects who have an initial TTP event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Time Frame: From treatment start date to date of progression/death, or censored as described; assessed for approximately 3 years.
Reporting Status: Not Posted, anticipated posting 2026-02

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR will be calculated for each subject with response for the VGPR+ and overall response endpoints. The DoR intervals will be calculated from the time of the first assessment that identified response until disease progression or death. The censoring mechanism for DoR will be the same as described for PFS.
Time Frame: From time of first response to date of progression/death, or censored as described; assessed for approximately 3 years.
Reporting Status: Not Posted, anticipated posting 2026-02

7. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT will be calculated from the time of treatment start until the start of the first subsequent anti-cancer therapy after all protocol directed therapy is completed. For surviving subjects who do not receiving subsequent therapy, TTNT will be censored at the last contact date. For subjects who die before beginning subsequent anti-cancer therapy, TTNT will be censored at the date of death
Time Frame: From treatment start date to date of next treatment, or censored as described; assessed for approximately 3 years.
Reporting Status: Not Posted, anticipated posting 2026-02

ADVERSE EVENTS:
Time Frame: Baseline, during treatment, and through 30 days after study treatment is discontinued, an average of 14 months.
Groups:
- KRd-Elotuzumab: Carfilzomib, Revlimid, Dexamethasone, Elotuzumab
  Elotuzumab: Experimental
Arm/Group | KRd-Elotuzumab
All-Cause Mortality (participants affected / at risk) | 6/15
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRd-Elotuzumab (N=15)
Anemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Fever (General disorders) | 6
Lung infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Renal Cell Carcinoma
Syncope (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hematoma (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRd-Elotuzumab (N=15)
Anemia (Blood and lymphatic system disorders) | 3
Cardiac disorders - Other (Cardiac disorders) | 1 — Cardiomegaly
Aortic Injury (Injury, poisoning and procedural complications) | 1
Cardiac disorders - Other (Cardiac disorders) | 1 — Elevated BNP
Aortic valve disease (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 2
Floaters (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 9
Edema limbs (General disorders) | 7
Pain (General disorders) | 5
Fever (General disorders) | 3
Injection site reaction (General disorders) | 1
Phlebitis (Vascular disorders) | 1
Chills (General disorders) | 1
Infusion related reaction (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 2
Bronchial infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 1 — Trichomonas
Lung infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 2
Cholesterol high (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 — Vitamin B12 deficiency
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Bunion, bilateral feet
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Cyst (L) posterior neck
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Top of L foot-no neoplasm
Headache (Nervous system disorders) | 7
Paresthesia (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 2
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 5
Agitation (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 — Dysuria
Urinary retention (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Skin open over PAC site
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Night sweats
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Hot sensation palms
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Scrape (L hand, R second toe)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 5
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 2
Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT03361306/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT03361306/ICF_001.pdf